CLINICAL TRIAL: NCT01344473
Title: A Randomised Controlled Trial of Tooth Mousse to Remineralise Post-orthodontic Treatment White Spot Lesions
Brief Title: A Trial of Tooth Mousse to Remineralise Post-orthodontic Treatment White Spot Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: NHS Tayside (Other Government)
Responsible Party: Principal Investigator, Fiona Hogarth, TCTU Assistant Director, University of Dundee
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010DE11; NCT01631734 (obsolete NCT alias)
Record Dates: First submitted 2011-04-07; First posted 2011-04-29 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Demineralisation; White Spot Lesions; Orthodontic Treatment
Keywords: Remineralisation; White Spot Lesions; Orthodontic treatment; Tooth Mousse creme; Casein Phosphopeptide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Casein phosphopeptide in the form of TM (Experimental): Experimental group will be given TM to use daily for 12 weeks
  Interventions: Device: Tooth Mousse creme (Casein Phosphopeptide)(RECALDENT)
- No intervention (No Intervention): Standard oral care

INTERVENTIONS:
Device: Tooth Mousse creme (Casein Phosphopeptide)(RECALDENT) — TM is a water based creme containing RECALDENT. RECALDENT consists of CPP-AP: Casein Phosphopeptide - Amorphous Calcium Phosphate.
  Other Names: RECALDENT
  Arms: Casein phosphopeptide in the form of TM

SUMMARY:
Fixed dental braces are associated with the risk of developing White Spot Lesions (WSLs), which appear as white chalky marks on the teeth. They develop as a result of the acid produced by bacteria in dental plaque dissolving the outer surface of the tooth, known as demineralisation. Recently, amorphous calcium phosphate (ACP) stabilised by casein phosphopeptide (CPP) has become available, and it is reported to help rebuild the surface of teeth which have WSLs. CPP-ACP is available incorporated into a crème known as Tooth Mousse (TM). While there appears to be sufficient evidence regarding the use of CPP-ACP in promoting general remineralisation, for the first time this study aims to examine the use of CPP-ACP to treat WSLs in post-orthodontic participants.

DETAILED DESCRIPTION:
The study will be run in the Orthodontic departments of Dundee Dental School and Perth Royal Infirmary, both in NHS Tayside. The investigators will recruit a total of 80 participants to the study. Clinicians within the orthodontic departments will determine when a patient could be a potential participant of the study, and one visit prior to debonding of their brace, the treating clinician will discuss the study with the potential participant. If they are interested in finding out more, the clinician will issue the potential participant with the appropriate PIL. There will be a PIL for potential participants over sixteen years old, and separate PILs for those aged twelve to sixteen years old, under twelve years old, and for parents/guardians of potential participants under sixteen years old.. The clinician will then inform the PI/SI that a PIL and supporting documentation has been issued. There will be a potential participant referral form, which can be completed to aid the transfer of information to the PI/SI. Potential participants under twelve years old will be advised that a parent or guardian must attend with them for the debond appointment, when written informed consent (IC) will be sought from the parents/guardians by the Investigators of the study.

Once IC has been obtained, resting and stimulated salivary flow rate will be measured by the Investigators or delegated member of the research team using a Saliva-Check Buffer kit (GC Corp, Leuven, Belgium). The kit will allow observation of the quantity and viscosity of resting saliva produced in one minute, and the pH of the sample will also be tested and recorded. Participants will then chew a piece of paraffin wax for a two-minute period to produce a stimulated salivary sample. The liquid component of the sample will be measured to allow a flow rate in ml/minute to be calculated, and the pH again tested and recorded. The buffering capacity of the stimulated saliva will also be determined by challenging the saliva with varying amounts of lactic acid. As a lack of saliva would bias the results for the study due to increased caries risk, and as saliva is essential for the hydrolysis of the CPP-ACP from the TM, if the resting salivary flow rate is below 0.2ml/min, or the stimulated rate below 1.0ml/min, then the subject will be excluded from the study. Participants will then be randomly allocated to the control or the experimental group.

Each subject included in the study will have their WSLs assessed and categorised clinically using the International Caries Detection and Assessment System, (ICDASii) (International Caries Detection and Assessment System Coordinating Committee, 2009a), by ICDASii calibrated examiners. Examiner reliability will be determined by scoring extracted teeth and teeth validated by histology. Reproducibility will be measured using Kappa scores. All lesions on the buccal surfaces of teeth will be included in the study. Intra-oral digital photographs will also be taken of each participant in a reproducible manner, and the photographs analysed by two different blinded ICDASii calibrated examiners, who will be recruited to the study simply to score the clinical photographs. A colour standard (CasMaTCH; Bear medic, Tokyo) will be used to allow colour matching of the images.

The experimental group will receive TM crème to use daily. The oral and written instructions regarding crème application will be provided, indicating that the crème should be applied to all surfaces of the teeth, agitated (swished) for one minute and then retainers placed for night-time wear as per crème application protocol.

Subjects in the control group will not use any crème in their retainers, but will simply be asked to place their retainer for night-time wear.

At commencement of the study it will be recorded how long participants fixed appliances had been in situ, and all participants and clinicians will receive a questionnaire to determine their fluoride use, oral hygiene regime, diet and preventive interventions e.g. visits to hygienist, topical fluoride application, during their fixed appliance treatment. The participants dental records will be reviewed and any record of pre-existing developmental defects of enamel or WSLs will be documented. Participants will be asked to score their own perception of the appearance of their teeth, considering the presence of their WSLs, using a validated Visual Analogue Scale (VAS).

Participants will be reviewed at 6 weeks and at 12 weeks. At both visits WSLs will be reassessed and categorised by a calibrated examiner (PI/SI) using ICDASii. Digital photographs will be retaken for analysis by other blinded, calibrated examiners and the where appropriate, the participants will be asked to bring their tube of unused crème to be weighed to help determine compliance to the study protocol. A decision has been made not to issue subject diaries to determine compliance as evidence in the Orthodontic literature hasn't found self-reporting of this type, in this area to be reliable. Participants will be asked to score the appearance of their teeth using the VAS again and subjects in the experimental group will complete a questionnaire on acceptability, taste and convenience of using the crème.

A transition matrix incorporating ICDASii severity and activity scores will be used to assess the stability, regression or progression of WSLs between baseline and follow-up examinations.

ELIGIBILITY:
Inclusion Criteria:

* Single or both arch fixed orthodontic appliance treatment completed
* Being provided with a vacuum formed retainer(s)
* Participant, or parent or guardian of participant if less than 12 years, gives written informed consent

Exclusion Criteria:

* Tooth Mousse used during orthodontic treatment
* Having a bonded retainer
* Not receiving a vacuum formed retainer
* Suffers from psychiatric or behavioural problems which may affect ability to follow study instructions
* Resting salivary flow rate less than 0.2ml/minute
* Stimulated salivary flow rate less than 1.0ml/minute
* Allergic to milk proteins or benzoate derivatives
* Unable to read and understand PIL, ICF and questionnaires
* Taking medication which may affect salivary flow

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-03; Primary Completion 2013-08 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Effectiveness of TM to promote remineralisation of WSLs | 12 weeks
  To determine the effectiveness of TM to promote remineralisation of WSLs in post orthodontic treatment study patients. Patients will be reviewed at 6 weeks and 12 weeks. At both visits WSLs will be reassessed and categorised by a calibrated examiner using the International Caries Detection and Assessment System (ICDASii) for scoring lesions. Examiner reliability will be determined by scoring extracted teeth and teeth validated by histology. Intra-oral photographs will also be taken of each participant and the photographs analysed by two different blinded ICDASii calibrated examiners.
Participants' perception of the appearance of their WSLs | 12 weeks
  To determine the change in study participants' perceptions of the appearance of their WSLs after using TM or no TM in their orthodontic retainers. Patients will be asked to score their own perception of the appearance of their teeth, considering the presence of their WSLs, using a Visual Analogue Score (VAS).

SECONDARY OUTCOMES:
Information on oral hygiene regimes and fluoride use during the period of fixed appliance treatment. | Week 0
  This outcome aims to obtain information on oral hygiene regimes and fluoride use during fixed appliance treatment of study participants who exhibit WSLs at the end of fixed appliance treatment. At the time of recruitment, it will be recorded how long participants' fixed appliances had been in situ and all participants and clinicians will receive a questionnaire to determine their fluoride use, oral hygiene regime, diet and preventive interventions e.g. visits to hygienist etc during their fixed appliance treatment.
Assess severity and location of WSLs in orthodontic treatment | Week 0
  At the time of recruitment, and immediatly after removal of their fixed appliance, the participants will have the severity and location of their WSLs assessed and categorised clinically using the ICDASii calibrated examiners. All lesions on the buccal surfaces of the teeth will be included in the study. Intra-oral digital photographs will also be taken of each participant and the photographs analysed by two different blinded ICDASii calibrated examiners.
Compare ICDASii scores in different assessment techniques | 12 weeks
  To compare the ICDASii scores of WSLs determined clinically with ICDASii scores of the same WSLs determined using digital photography 6 weeks and 12 weeks after debond of their appliance.

CONTACTS AND LOCATIONS:
Overall Officials: David Bearn, M(Orth)RCS PhD BDS, Principal Investigator — University of Dundee; Louise Greene, MFDS BDS, Principal Investigator — NHS Tayside
Locations (2):
- United Kingdom (2):
  - Dundee Dental Hospital, Dundee
  - Perth Royal Infirmary, Perth

REFERENCES:
- [Background] Manton DJ, Shen P, Cai F, Cochrane NJ, Reynolds C, Messer LB, Reynolds EC. Remineralisation of WSLs in situ by TM. (Abstract) IADR 84th General Session, Brisbane 2006.
- [Background] Morgan MV, Bailey D, Adams G, Tsao C, Hyslop A, Escobar K, Manton DJ, Reynolds E. A clinical study measuring white spot lesion progression and regression. (Abstract) J Dent Res 2008: 87 (special issue B): 11-4